CLINICAL TRIAL: NCT03358589
Title: Molecular Evaluation in Metastatic Breast Cancer - A Clinical Study of Accuracy and Response Assessment
Brief Title: Molecular Evaluation in Metastatic Breast Cancer
Acronym: MESTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Vogsen, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MESTAR
Record Dates: First submitted 2017-11-09; First posted 2017-11-30 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Breast Cancer; Molecular Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Masking Description: it is a single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MESTAR (Other): All patients will have the same scans performed
  Interventions: Diagnostic Test: FDG-PET/CT

INTERVENTIONS:
Diagnostic Test: FDG-PET/CT — Scans
  Other Names: WBMRI

SUMMARY:
Background: Despite that up 90% of patients with early-stage breast cancer receives adjuvant treatment, there are still about 300 patients diagnosed with primary metastatic breast cancer (MBC) and about 1,200 patients who develop metastases after the primary treatment each year in Denmark.

Aim: The investigators hypothesize that molecular evaluation with FDG-PET/CT and diffusion weighted MRI allows an earlier detection of failure to respond to potentially toxic drugs in patients receiving breast cancer directed treatments.

The aims of our project are to address the following questions:

* Does FDG-PET/CT allow an earlier detection of failure to respond to treatment for MBC than conventional CT?
* Does FDG-PET/CT or MRI allow an earlier detection of failure to respond to treatment for bone metastatic disease than conventional CT?
* Does the PET based criteria (PERCIST) have the potential to lead to changes in the treatment plans made from CT based criteria (RECIST)?
* Does FDG-PET/CT give a more accurate diagnosis of MBC than conventional CT in terms of number and distribution of metastatic sites?

Method: Part A - the accuracy study: The study population will comprise all women referred to Odense University Hospital with suspected metastatic breast cancer (MBC). The investigators expect to include 270 patients who will be examined with FDG-PET/CT. If bone metastases are detected, the patients will proceed to MRI. All patients with suspected metastases on FDG-PET/CT or MRI will have a biopsy from a suitable lesion Part B - the response evaluation study: The investigators expect to include 90 patients with biopsy-verified MBC. Patients will receive oncologic treatment according to national guidelines. Response to treatment will be evaluated by conventional CT criteria and compared to novel criteria according to FDG- PET/CT, and MRI. Test results will be blinded to each other, so that knowledge of other test results will be unknown for the reader of the CT, FDG-PET/CT or MRI, respectively Expected clinical impact: This project represents a truly multidisciplinary effort to improve the diagnosis, staging, and response evaluation of MBC. The investigators hope that patients will benefit in terms of being spared for ineffective toxic treatment due to earlier detection of failure to respond, and hence leading to earlier treatment transition. Patients are involved in the planning and conduct of the project.

DETAILED DESCRIPTION:
Background Breast cancer is the most frequent malignant disease in Danish women with about 4,500 new cases per year and about 60,000 women living after a diagnosis of breast cancer (1). After lung cancer, it is the most common cause of death from cancer among Danish women. Despite that up 90% of patients with early-stage breast cancer receive adjuvant treatment, there are still about 300 patients diagnosed with primary metastatic breast cancer and about 1,200 patients who develop metastases after the primary treatment each year in Denmark (2). Clinical guidelines unanimously recommend that diagnostic work-up for metastatic disease should be performed only when clinically indicated, or prior to primary treatment in patients at high risk of MBC, but they do not make clear recommendations on which diagnostic tool to apply for staging patients with suspected MBC (3-5). The investigators have shown recently that the molecular whole body imaging with FDG-PET/CT has a higher accuracy than conventional imaging with CT and bone scintigraphy when diagnosing MBC (6); the investigators results are in accordance with existing meta-analyses (7,8), and a recent review (9).The gold standard for verifying MBC is a biopsy from a metastatic lesion, but treatment decisions are often based on the biomarker profile of the primary tumor, since it has been assumed to remain the same in the corresponding metastatic lesions. The investigators own data (10) supported by a meta-analysis (11) point towards discordances between the primary tumor and the corresponding metastasis ranging from 9% to 23% for expression of estrogen receptors (ER), Human Epidermal growth factor receptor 2 (HER-2), and Topoisomerase 2A (TOP2A).

It is essential to know the exact baseline stage of MBC in order to allow adequate evaluation of treatment response subsequently. Response evaluation criteria have traditionally been based on the morphological size of solid tumors as in the Response Evaluation Criteria in Solid Tumors (RECIST)(12). The investigators consider it important to include changes in metabolic activity for evaluation of treatment response, since metabolic changes occur before morphological changes can be detected. The PET response Criteria in Solid Tumors (PERCIST) is a new standardized method to assess quantitatively the metabolic tumor response as seen on FDG-PET/CT (13). A recent pooled analysis and review comparing the PERCIST to the RECIST criteria concluded that the PERCIST criteria seem to be more suitable for assessing tumor response than the RECIST criteria, but that the role of the PERCIST criteria needs to be validated in relevant clinical settings (14).

Monitoring response to therapy in skeletal metastases has been challenging because the RECIST criteria do not include changes in bony structures though the RECIST 1.1 accepts bone metastases with soft tissue masses measuring >= 10 mm as a target lesion (15). Up to 70% of patients with MBC present with bone involvement, characterized as osteolytic, osteoblastic, or mixed lesions on CT. Soft tissue metastases in the bone marrow may be overlooked by conventional imaging, but magnetic resonance imaging (MRI) has shown high accuracy for diagnosing bone and bone marrow metastases (16, 17). Molecular imaging with FDG-PET/CT and diffusion weighted MRI both have the potential to detect metabolic activity in all types of bone and bone marrow lesions, and therefore a combination of FDG-PET/CT and whole body MRI (WBMRI) may give valuable information in assessing metastatic processes in bone.

Aim The investigators hypothesize that

•Molecular evaluation can provide a more accurate assessment of the metastatic spread than conventional methods and that molecular evaluation of response to breast cancer directed treatments allows an earlier detection of failure to respond to potentially toxic drugs.

The aims of the project are to address the following questions:

* Does FDG-PET/CT allow an earlier detection of failure to respond to treatment for MBC than conventional CT?
* Does FDG-PET/CT or MRI allow an earlier detection of failure to respond to treatment for bone metastatic disease than conventional CT?
* Does the PET based criteria (PERCIST) have the potential to lead to changes in the treatment plans made from CT based criteria (RECIST)?
* Does FDG-PET/CT give a more accurate diagnosis of MBC than conventional CT in terms of number and distribution of metastatic sites?

Method The project is divided into 2 parts. Part A - the accuracy study: The study population will comprise all women referred to Odense University Hospital (OUH) with a suspected first recurrence of breast cancer and newly diagnosed breast cancer at high risk of metastatic spread. Data will be collected from about 270 patients over a 2-year period (Figure 1) All patients will be examined by FDG- PET/CT with contrast enhanced CT in diagnostic quality at baseline. If bone metastases are detected, the patients will proceed to WBMRI. All patients with suspected metastases on FDG-PET/CT or WBMRI will have a biopsy from a suitable lesion. The tissue from the biopsy will be for standard diagnostic procedures, including immunohistochemistry for biomarkers (ER, HER-2).

All non- metastatic patients will be followed for one year by medical records to detect potentially false negatives.

Part B - the response evaluation study: The response evaluation part is planned as a longitudinal cohort design analyzing change of management and prediction og progression free survival. It will include about 90 patients expected to present with biopsy-verified MBC during the inclusion period. (Figure 1).

Patients will receive oncologic treatment directed by the biomarker profile of the biopsy and according to national guidelines. Response to treatment will be evaluated by FDG-PET/CT with contrast enhanced CT in diagnostic quality after three series of chemotherapy (every 9 weeks) or after 3 months of endocrine therapy (every 12 weeks). Patients with bone metastases will be evaluated by WBMRI as well. Lesion based sensitivity analyses will be made for FDG-PET/CT and for diagnostic CT, and in patients with bone involvement also for WBMRI. A radiologist will apply the RECIST criteria from the CT and dedicated diffusion measurements from the MRI, while a Nuclear Medicine Physician will apply the PERCIST criteria along with other relevant quantitative measures. Test results will be blinded to each other, so that knowledge of other test results will be unknown for the reader of the CT, FDG-PET/CT or MRI, respectively. Treatment decisions will be made in a multidisciplinary conference form. Decisions will be based on the conventional imaging criteria (RECIST) in the first 30 patients, and for each patient the decision will be reconsidered by the PERCIST criteria and the metabolic measurements. Discrepancies in decisions guided by the different evaluation criteria will be registered and analyzed with regard to change of management in an interim analysis. The same will be done for the succeeding evaluations, but the choice of response evaluation criteria to guide clinical decision will depend on the result of the interim analysis.

The investigators plan the data collection in a way that allows us to perform cost-effectiveness analyses for the response evaluation study.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age > 18
* Suspicion of recurrence of earlier breast cancer or new breast cancer diagnose with high risk of metastatic disease
* Life expectancy > 3 month
* Signed statement of consent

Exclusion Criteria:

* Men
* Pregnancy
* Severe Medical conditions
* severe mental og psychological conditions
* contraindications for MRI (for patients with bone metastasis)
* treatment for other malignant diseases within the last 5 years prior to inclusion (except carcinoma in situ cervicis uteri and basal cell carcinoma (BCC))

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to breast cancer. Rare among men
Enrollment: 270 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  Lesion based sensitivity analyses will be made for FDG-PET/CT and for diagnostic CT, and in patients with bone involvement also for WBMRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Marianne Vogsen, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogsen M, Naghavi-Behzad M, Harbo FG, Jakobsen NM, Gerke O, Asmussen JT, Nissen HJ, Dahlsgaard-Wallenius SE, Braad PE, Jensen JD, Ewertz M, Hildebrandt MG. 2-[18F]FDG-PET/CT is a better predictor of survival than conventional CT: a prospective study of response monitoring in metastatic breast cancer. Sci Rep. 2023 Apr 5;13(1):5552. doi: 10.1038/s41598-023-32727-w. PMID 37019987
- [Derived] Vogsen M, Jensen JD, Gerke O, Jylling AMB, Asmussen JT, Christensen IY, Braad PE, Thye-Ronn P, Soe KL, Ewertz M, Hildebrandt MG. Benefits and harms of implementing [18F]FDG-PET/CT for diagnosing recurrent breast cancer: a prospective clinical study. EJNMMI Res. 2021 Sep 22;11(1):93. doi: 10.1186/s13550-021-00833-3. PMID 34553294
- [Derived] Vogsen M, Geneser S, Rasmussen ML, Horder M, Hildebrandt MG. Learning from patient involvement in a clinical study analyzing PET/CT in women with advanced breast cancer. Res Involv Engagem. 2020 Jan 6;6:1. doi: 10.1186/s40900-019-0174-y. eCollection 2020. PMID 31921443